CLINICAL TRIAL: NCT00707174
Title: Combination Therapy With Imiquimod Cream 5% and Tazarotene Cream 0.1% for the Treatment of Lentigo Maligna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI13361
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Cancer; Lentigo Maligna
Keywords: Lentigo Maligna
MeSH Terms: conditions — Neoplasms; Hutchinson's Melanotic Freckle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Topical imiquimod group:
  treat the LM site two centimeters beyond the perimeter margin with topical imiquimod 5% cream Monday thru Friday of each week for a total of twelve weeks. After three months of topical treatment, a one-month wash out period will be observed to allow for resolution of inflammation that can obscure the pathologist's ability to evaluate the excised tumor/treatment site.
  Interventions: Drug: Imiquimod Cream
- 2 (Experimental): Topical imiquimod and topical tazarotene 0.1% cream group:
  Patients randomized to this group will undergo an identical treatment protocol as the topical imiquimod group with the addition of topical tazarotene 0.1% cream on Saturday and Sunday of each week.
  Interventions: Drug: Tazarotene Cream 0.1%

INTERVENTIONS:
Drug: Imiquimod Cream — Our current standard-of-care is to use imiquimod daily for 12 weeks followed by a staged-excision with 2mm margins per stage. These margins are justified because the standard-of care for lentigo maligna is continuing to evolve
  Arms: 1
Drug: Tazarotene Cream 0.1% — Tazarotene is a topical retinoid cream that is commonly used to treat psoriasis and acne. It is known to help keratinocyte maturation and thinning of the stratum corneum (top layer of the epidermis). The stratum corneum functions as the primary barrier to the penetration of topical medications. The penetration of topical medications can be enhanced if the stratum corneum is thinned. We believe that the treatment of lentigo maligna with imiquimod, and staged-excision, will be improved by the addition of tazarotene cream.
  Arms: 2

SUMMARY:
This study is designed as a randomized, prospective study to test the efficacy of imiquimod plus tazarotene in the treatment of LM. Eligible and consented patients will be randomized to one of two treatment groups: 1) topical imiquimod group, or 2) topical imiquimod combined with topical tazarotene group. All patients will undergo a staged surgical excision with rush permanent sections to confirm negative histologic margins. This will be followed by a surgical repair of the defect and long-term follow-up of five years to rule out recurrences. Both groups will have a polygonal excision using 2mm margins per stage.

DETAILED DESCRIPTION:
Objectives

The objectives of the study are:

1. reduce the surgical morbidity of staged excisions which often require multiple stages of surgery in order to verify negative histologic margins
2. investigate the addition of a topical retinoid, to our standard-of-care (topical imiquimod and staged-excision) and evaluate if there is improvement in efficacy
3. to see if treatment of surrounding normal appearing skin with this combination of topical agents reduces recurrence rates compared to staged-excision. Our hypothesis is that the combination of topical agents will better treat the subclinical melanocytic atypia which can give rise to recurrences.

Primary endpoint:

The primary goal is a comparison of the number of stages required for negative histologic margins in the imiquimod plus tazarotene group compared to the imiquimod group. Tumors requiring 5 or more stages in will be combined into one category for data analysis. The Wilcoxon-Mann-Whitney test will be used for statistical comparison.

Secondary endpoints:

1. Comparison of the surgical defect size (mm2) between the study groups. The difference in area between the entire surgical defect and the original tumor (as recorded on transparent plastic) will be calculated for each patient and used as an endpoint.
2. Comparison of skin inflammation between the study groups. Skin inflammation will be recorded as an ordered categorical variable with four categories (0-3) as described in Section 5.
3. The type of surgical repair required (i.e. primary repair, skin flap, skin graft).
4. Immunostaining to evaluate inflammatory infiltrate. Immunostaining will be analyzed as an ordered categorical variable.
5. Recurrence of the tumor at 3 months, 6 months, 12 months, and yearly for the next four years.
6. The proportion of patients with skin ulceration.
7. The relationship between ulceration, skin inflammation and clearance of LM.

Study Procedures A total of eighty patients, over a twelve-month period, will be recruited from one center for this open label study. Forty patients will be randomly assigned to one of two treatment groups as mentioned in the Study Design section. The study will consist of 4 phases: (1) Enrollment and screening period to evaluate skin cancer, measure and trace its perimeter; (2) 12 week treatment with topical application of study drug(s); (3) Surgical excision of treatment site to ensure eradication of the tumor; (4) Follow-up period to rule out recurrences.

All patients must have a biopsy-proven diagnosis of lentigo maligna confirmed by at least two dermatopathologists from the Department of Dermatology at the University of Utah School of Medicine. At the initial examination the clinical borders of the lesion will be defined using a Wood's lamp (360nm) and the perimeter will be outlined with a gentian violet marker and photographed for the medical record. (Wood's lamp examination helps to identify pigmentary alterations of the skin when are sometimes difficult to appreciate under normal lighting conditions.) At the time of enrollment, to rule out an invasive melanoma, all potential study participants will undergo a shave biopsy of their lesion using local anesthesia. Enrollment will not occur until the biopsy has been examined and confirmed to be a lentigo maligna (melanoma in-situ). If an invasive melanoma is found, the patient will be excluded from the study and additional evaluation/therapies implemented. If the patient is enrolled in the study, a piece of their biopsy specimen will be used to perform immunohistochemistry to evaluate the inflammatory infiltrate. A similar series of histochemical staining will be performed at the conclusion of the study using a piece of the excised skin.

Topical imiquimod group:

Patients randomized to this group will have the perimeter of the LM site, as defined by a Wood's lamp examination, drawn on the skin with a gentian violet pen and photographed with a Polaroid camera . One photograph will go to the medical record and the second given to the patient to help identify the proposed treatment area. The gentian violet perimeter will then be copied on transparent plastic to facilitate tumor localization since the tumor is predicted to disappear clinically during treatment. The patients will then treat the LM site two centimeters beyond the perimeter margin with topical imiquimod 5% cream Monday thru Friday of each week for a total of twelve weeks. After three months of topical treatment, a one-month wash out period will be observed to allow for resolution of inflammation that can obscure the pathologist's ability to evaluate the excised tumor/treatment site. A staged excision will then be performed with two millimeter margins around the original tumor perimeter as previously recorded on transparent plastic which will be placed on the patient's skin to outline the perimeter accurately. Once negative margins are confirmed histologically, post-operative defect size will be measured in mm2 and then a plastic surgical repair will be performed to optimize cosmesis.

Topical imiquimod and topical tazarotene 0.1% cream group:

Patients randomized to this group will undergo an identical treatment protocol as the topical imiquimod group with the addition of topical tazarotene 0.1% cream on Saturday and Sunday of each week.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of eighty subjects who are 18 years or older and have a biopsy-proven lentigo maligna.
* The subjects must have a LM that is in a location amenable to treatment with imiquimod, express a willingness and ability to comply with study requirements, and tolerate an outpatient surgical procedure.
* All participants will sign consent documents prior to enrollment.
* The typical age of patient that develops a LM is beyond the child-bearing range.

Exclusion Criteria:

* In the event that a patient with a LM is pregnant, they will be excluded from the study.
* inability to tolerate the surgical procedure
* invasive melanoma
* previous surgery on the site of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Bowen, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Hyde MA, Hadley ML, Tristani-Firouzi P, Goldgar D, Bowen GM. A randomized trial of the off-label use of imiquimod, 5%, cream with vs without tazarotene, 0.1%, gel for the treatment of lentigo maligna, followed by conservative staged excisions. Arch Dermatol. 2012 May;148(5):592-6. doi: 10.1001/archdermatol.2012.270. PMID 22431716
- [Derived] Ho PA, Kopecky KJ, Alonzo TA, Gerbing RB, Miller KL, Kuhn J, Zeng R, Ries RE, Raimondi SC, Hirsch BA, Oehler V, Hurwitz CA, Franklin JL, Gamis AS, Petersdorf SH, Anderson JE, Godwin JE, Reaman GH, Willman CL, Bernstein ID, Radich JP, Appelbaum FR, Stirewalt DL, Meshinchi S. Prognostic implications of the IDH1 synonymous SNP rs11554137 in pediatric and adult AML: a report from the Children's Oncology Group and SWOG. Blood. 2011 Oct 27;118(17):4561-6. doi: 10.1182/blood-2011-04-348888. Epub 2011 Aug 26. PMID 21873548

RESULTS

PARTICIPANT FLOW:
Groups:
- Imiquimod Only: Topical imiquimod group:
  treat the LM site two centimeters beyond the perimeter margin with topical imiquimod 5% cream Monday thru Friday of each week for a total of twelve weeks. After three months of topical treatment, a one-month wash out period will be observed to allow for resolution of inflammation that can obscure the pathologist's ability to evaluate the excised tumor/treatment site.
- Imiquimod and Tazarotene Combined: Topical imiquimod and topical tazarotene 0.1% cream group:
  Patients randomized to this group will undergo an identical treatment protocol as the topical imiquimod group with the addition of topical tazarotene 0.1% cream on Saturday and Sunday of each week.
Period: Overall Study
Arm/Group | Imiquimod Only | Imiquimod and Tazarotene Combined
Started | 46 | 44
Completed | 41 | 37
Not Completed | 5 | 7
Not completed — Adverse Event | 1 | 6
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imiquimod Only | Imiquimod and Tazarotene Combined | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 16 | 37
  >=65 years | 25 | 28 | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 67.87234 (13.07606) | 67.40909 (11.99286) | 67.64 (12.49655)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 35 | 31 | 66
Region of Enrollment [Number; unit: participants]
  United States | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: The Absence of Lentigo Maligna (LM) at the Time of Staged Excisions in Participants
Description: Negative histologic margins for the imiquimod plus tazarotene group compared to the imiquimod only group.
Time Frame: 24 months
Population: All evaluable patients from both groups were compared
Measure: Number; unit: participants
Arm/Group | Imiquimod Only | Imiquimod and Tazarotene Combined
Number analyzed (Participants) | 41 | 37
participants | 27 | 29

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Imiquimod Only | Imiquimod and Tazarotene Combined
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 1/46 | 6/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod Only (N=46) | Imiquimod and Tazarotene Combined (N=44)
Inflammatory Response (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes